CLINICAL TRIAL: NCT05610215
Title: Concomitant Hybrid Versus Catheter Ablation for Reinforcing Therapeutic Effect of Atrial Fibrillation With Hypertrophic Cardiomyopathy
Brief Title: Concomitant Hybrid Versus Catheter Ablation for Atrial Fibrillation With Hypertrophic Cardiomyopathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-1736
Record Dates: First submitted 2022-11-02; First posted 2022-11-09 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Atrial Fibrillation; Cardiomyopathy, Hypertrophic; Radiofrequency Ablation
MeSH Terms: conditions — Atrial Fibrillation; Cardiomyopathy, Hypertrophic | interventions — Catheter Ablation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hybrid ablation (Experimental): Participants in this group will receive concomitant thoracoscopic epicardial ablation and catheter endocardial ablation
  Interventions: Procedure: hybrid ablation
- catheter ablation (Active Comparator): Participants in this group will receive catheter endocardial ablation only
  Interventions: Procedure: catheter ablation

INTERVENTIONS:
Procedure: hybrid ablation — simultaneous thoracoscopic epicardial and catheter endocardial ablation
  Arms: hybrid ablation
Procedure: catheter ablation — catheter endocardial ablation
  Arms: catheter ablation

SUMMARY:
The goal of this clinical trial is to compare the rhythm control effect in hypertrophic non-obstructive patients with non-paroxysmal atrial fibrillation by either concomitant catheter endocardial and thoracoscopic epicardial ablation or catheter ablation alone. The study aims to see if concomitant hybrid ablation can more effectively achieve rhythm control effect than catheter ablation alone in non-paroxysmal atrial fibrillation patients with hypertrophic cardiomyopathy.

DETAILED DESCRIPTION:
After informed consent, 66 eligible admissions will be recruited in 2 centers. Eligible participants will be randomly divided (1:1) into either hybrid or catheter ablation arms, looking for a primary outcome of 1-year freedom from atrial arrhythmias.

ELIGIBILITY:
Inclusion Criteria:

1. Patients' age is ≥18 y
2. Clinically diagnosed hypertrophic cardiomyopathy (any left ventricular wall segment thickness ≥15 mm in genetical negative (or unknown genetical status) patients or ≥13mm in genetical positive ones-as measured by any imaging technique (echocardiography, cardiac magnetic resonance imaging or computed tomography)-that is not explained solely by loading conditions)
3. Non-obstructed left ventricular outflow obstruction with peak gradients <30mmHg
4. Concomitant with persistent atrial fibrillation (7 days<sustained episode lasting<3 years) with drug-refractory symptoms.
5. Be able to understand the contents of the trial, and provide written informed consent to participate in this investigation.

Exclusion Criteria:

1. Patients with left atrial size >60 mm (2-dimensional echocardiography, parasternal long-axis view)
2. Contraindicated to systemic anticoagulation
3. Left ventricular ejection fraction ≤40%
4. Concomitant with left atrium or left atrial appendage emboli
5. Concomitant with a coronary or valvular disease that indicates intervention
6. Ischaemic stroke within 2 months
7. Previous ablation history
8. Uncontrolled hyper/hypothyroidism
9. End-staged kidney failure
10. Concomitantly involved in other trials
11. Pregnant or breastfeeding, or women of childbearing age not using a reliable contraceptive method
12. Concomitant with bacteremia or at an active phase of infection
13. Anatomically not suitable for thoracoscopic surgery(history of chest surgery or radiotherapy, etc.)
14. Unwilling or unable to comply with all peri-ablation and follow-up requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-02-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Freedom from documented recurrence (off-AADs) | within 3-12 months
  freedom from documented AF/AT episodes >30 seconds (off-AADs) by 72-hour holter monitoring

SECONDARY OUTCOMES:
All cause mortality | within 12 months
  death by any reason
Cardiovascular related mortality | within 12 months
  death that related to cardiogenic causes
Cerebral infarction/ischemia | within 12 months
  Any stroke or TIA diagnosed in the clinical record after the completion of the intervention
Periferal arterial embolism | within 12 months
  Periferal arterial embolism
All-cause rehospitalization | within 3-12 months
  Rehospitalized by any reason
Heart failure related rehospitalization | within 3-12 months
  Rehospitalized by the cause of heart failure episode
Freedom from documented recurrence (on-AADs) | within 3-12 months
  freedom from documented AF/AT episodes >30 seconds (on-AADs) by 72-hour holter monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Zhe Zheng, MD.PhD, Study Chair — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai Hospital, National Center for Cardiovascular Diseases, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China

REFERENCES:
- [Derived] Tang Y, Li L, Chen S, Xue Y, Guo H, Song L, Tang M, Yao Y, Zheng Z. Hybrid versus catheter ablation for Hypertrophic CardioMyopathy with Atrial Fibrillation (HCM-AF): study protocol for a randomised controlled trial. BMJ Open. 2024 Oct 9;14(10):e089284. doi: 10.1136/bmjopen-2024-089284. PMID 39384237